CLINICAL TRIAL: NCT02609035
Title: Immunization Services Model for Adult Rate Improvement
Acronym: ImmuSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacy Quality Alliance (Other)
Responsible Party: Principal Investigator, Samuel Stolpe, Senior Director, Quality Strategies, Pharmacy Quality Alliance
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00014163
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Pharmacy; Immunization; Vaccines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients who are either appointment-based medication synchronization calls, refill ready calls, or refill reminder calls at the pharmacy who have been identified as missing at least one vaccination. These patients will receive a telephonic prompt to get a vaccination.
  Interventions: Behavioral: Telephonic prompt
- Control (No Intervention): Patients who are either appointment-based medication synchronization calls, refill ready calls, or refill reminder calls at the pharmacy who have been identified as missing at least one vaccination. These patients will receive usual pharmacy care.

INTERVENTIONS:
Behavioral: Telephonic prompt
  Other Names: Appended message
  Arms: Intervention

SUMMARY:
ImmuSMART is a study of personalized telephonic prompts to community pharmacy patients to improve adult vaccination rates for pneumococcal and herpes zoster vaccines.

DETAILED DESCRIPTION:
This study will investigate immunization rate improvement among adult patients in 250 northeastern US community pharmacies as a result of telephonic prompts during regular automated outbound communiqués. There will be three projects assessing different forms of these appended prompts-appointment-based medication synchronization automated prompts, refill ready automated prompts, and refill reminder automated prompts. Each intervention will occur in one of three pharmacy chains, each with approximately 10,000 patients randomized to control or intervention (receive prompt or no).

Prior to the outbound automated call to the patient, a third-party technology vendor (Scientific Technologies Corporation) will perform an automated immunization status assessment of the patient by submitting a query the state immunization registry to compare the adult patient's existing immunization record to the CDC Recommended Adult Immunization Schedule. Gaps in immunizations that fall within pharmacy scope of practice will be identified. During the automated call (performed by VoicePort, a pharmacy telephonic support vendor) to the patient, they will be prompted to receive identified immunization gap vaccines upon their next pharmacy visit, with priority on pneumococcal, influenza, and herpes zoster vaccinations. If the patient accepts, the vaccination will be delivered when next the patient comes to visit the pharmacy.

After 6 months of running the trial, statistical modeling will be employed to assess vaccination rate differences between control and intervention patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 19 years of age at date of enrollment
* Patient not in long-term care, hospice or otherwise identified as unable to come to pharmacy for receipt of vaccine
* Patient currently missing a record of receipt of at least one of three vaccinations: flu, pneumonia, or shingles
* Patient enrolled in telephonic pharmacy reminder service

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22301 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Vaccination rates | 3 months
  Administration of vaccine will be assessed at 3 months after patient receives the prompt